CLINICAL TRIAL: NCT03318783
Title: Subarachnoid Hemorrhage and Soluble Epoxide Hydrolase Inhibition Trial
Acronym: SUSHI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Ross Martini, MD, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17614
Record Dates: First submitted 2017-10-10; First posted 2017-10-24 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Delayed Cerebral Ischemia; Vasospasm, Cerebral; Endothelial Dysfunction
Keywords: Eicosanoids; Epoxyeicosatrienoic Acids
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — N-((4-cyano-2-(trifluoromethyl)phenyl)methyl)-3-((4-methyl-6-(methylamino)-1,3,5-triazin-2-yl)amino)cyclohexanecarboxamide

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of the two treatment arms based on an unrestricted or "fair-coin" randomization procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational pharmacy staff will maintain the randomization list and study/drug placebo assignment. Participants, care providers, the investigators and outcomes assessors will be blinded to the grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK2256294 (Active Comparator): 10mg capsules of GSK2256294 will be administered in a single dose once daily enterally for a duration of 10 days.
  Interventions: Drug: GSK2256294
- Placebo (Placebo Comparator): 10mg matched placebo capsules will be administered in a single dose once daily enterally for a duration of 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2256294 — GSK2256294 will be administered in a single dose once daily enteral for a duration of 10 days.
  Arms: GSK2256294
Drug: Placebo — Placebo will be administered in a single dose once daily enteral for a duration of 10 days.
  Arms: Placebo

SUMMARY:
Soluble epoxide hydrolase (sEH) is the metabolizing enzyme of epoxyeicosatrienoic acids (EETs), which may play a role in reducing neuroinflammation and regulating cerebral blood flow after subarachnoid hemorrhage (SAH). Hypotheses: Pharmacologic inhibition of the sEH enzyme is safe and will result in increased EETs availability in the blood and cerebrospinal fluid. This study is a double-blind, placebo-controlled, phase 1b randomized trial to evaluate the safety and efficacy of GSK2256294, a novel soluble epoxide hydrolase inhibitor in patients with aneurysmal SAH.

DETAILED DESCRIPTION:
Study Description: Soluble epoxide hydrolase (sEH) is the metabolizing enzyme of epoxyeicosatrienoic acids (EETs), which may play a role in reducing neuroinflammation and regulating cerebral blood flow after subarachnoid hemorrhage (SAH).

Hypothesis: Pharmacologic inhibition of the sEH enzyme is safe and will result in increased EETs availability at the neurovascular unit, and a measured increase in the EET/DHET ratio in the serum and cerebrospinal fluid. This study is a double-blind, placebo-controlled, phase 1b randomized trial to evaluate the safety and of GSK2256294, an inhibitor of soluble epoxide hydrolase, in patients with aneurysmal SAH.

Objectives:

Primary Objective:

Determine the safety of administration of GSK2256294 in patients with aneurysmal SAH.

Secondary Objective:

Determine the pharmacodynamic effect of administration of GSK2256294 in patients with aneurysmal SAH on reducing EETs metabolism and biomarkers of cerebrovascular inflammation and endothelial injury.

Tertiary Objective:

Provide preliminary estimates of clinical endpoints to inform the design of a larger trial

Endpoints:

Primary Endpoints:

Determination of safety

Secondary endpoints:

1. Study days 7 and 10 serum EET/DHET ratios
2. Study days 7 and 10 cerebrospinal fluid (CSF) EET/DHET ratios
3. Study days 7 and 10 serum EPOME/DPOME ratio
4. Neuroinflammatory and endothelial injury biomarker levels from the blood and CSF at day 7 and day 10.

Tertiary, exploratory endpoints:

Clinical outcomes associated with SAH including neurologic status, disposition, vital status and incidence of delayed cerebral ischemia.

20 subjects will be randomized. Patients age 18 or above with confirmed ruptured aneurysms will be approached to provide written informed consent

Phase: Phase 1B

Description of Sites/Facilities Enrolling Participants: The study will take place at Oregon Health & Science University Hospital, with enrollment of patients admitted to the OHSU NSICU, a part of a comprehensive stroke center certified by the American Heart Association and Joint Commission for Accreditation of Healthcare Organizations, with a catchment area including the state of Oregon, Southwest Washington and Northern California. Approximately 80-100 patients with aneurysmal SAH are admitted each year.

Description of Study Intervention: Twenty patients will be equally randomized to receive once daily either 10 mg dose of GSK2256294 or placebo enterally for a duration of 10 days.

Study Duration: 24 months

Participant Duration: 90 days

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Head CT evidence of subarachnoid hemorrhage
3. Digital subtraction cerebral angiography or CT angiogram documenting the presence of a cerebral aneurysm.

Exclusion Criteria:

1. Symptom onset compatible with SAH of > 3 days prior to admission to OHSU
2. Absence of an indwelling external ventricular drain
3. Administration of any of the following inducers/inhibitors of CYP3A4: ritonavir, indinavir, nelfinavir, saquinavir, clarithromycin, telithromycin, chloramphenicol, ketoconazole, itraconazole, nefazodone, cobicistat or enzalutamide.
4. Suspected or confirmed pregnancy
5. Preexisting severe neurologic deficit or condition
6. Chronic renal failure requiring dialysis
7. Severe terminal disease with life expectancy <6 months
8. Unable to read or understand written or spoken English or Spanish
9. Refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Martini, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Martini RP, Siler D, Cetas J, Alkayed NJ, Allen E, Treggiari MM. A Double-Blind, Randomized, Placebo-Controlled Trial of Soluble Epoxide Hydrolase Inhibition in Patients with Aneurysmal Subarachnoid Hemorrhage. Neurocrit Care. 2022 Jun;36(3):905-915. doi: 10.1007/s12028-021-01398-8. Epub 2021 Dec 6. PMID 34873674

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2256294 | Placebo
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 subject in the placebo group died on study day 9 after having received 9 of 10 doses of study drug. Data is included for this subject throughout the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2256294 | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.2) | 60.4 (11.4) | 60.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (6.6) | 27.7 (4.7) | 28.2 (5.6)
Smoking [Count of Participants; unit: Participants]
  Never/Passive Smoker | 2 | 5 | 7
  Active Smoker | 5 | 3 | 8
  Former Smoker | 3 | 1 | 4
History of Hypertension [Count of Participants; unit: Participants] | 6 | 9 | 15
History of Seizure [Count of Participants; unit: Participants] | 0 | 0 | 0
History of Prior Brain Aneurysm [Count of Participants; unit: Participants] | 1 | 0 | 1
Pre-Admission Antihypertensives [Count of Participants; unit: Participants] | 3 | 8 | 11
Pre-Admission Anticoagulants [Count of Participants; unit: Participants] | 0 | 2 | 2
Pre-Admission Antiplatelet Agents [Count of Participants; unit: Participants] | 2 | 2 | 4
Pre-Admission Statins [Count of Participants; unit: Participants] | 1 | 1 | 2
Pre-Admission Antidiabetic Agents [Count of Participants; unit: Participants] | 0 | 0 | 0
Hunt and Hess Scale [Mean (Standard Deviation); unit: units on a scale] — The Hunt and Hess scale is a grading system used to classify the severity of a subarachnoid hemorrhage based on the patient's clinical condition.
  Description:
  1. - Asymptomatic, mild headache, slight nuchal rigidity
  2. - Moderate to severe headache, nuchal rigidity, no neurologic deficit other than cranial nerve palsy
  3. - Drowsiness / confusion, mild focal neurologic deficit
  4. - Stupor, moderate-severe hemiparesis
  5. - Coma, decerebrate posturing
  units on a scale | 3.0 (.94) | 3.0 (1.0) | 3.0 (.94)
Modified Fisher Grade [Mean (Standard Deviation); unit: units on a scale] — The modified Fisher scale is a method for grading subarachnoid hemorrhage (SAH) severity seen on non-contrast CT. The risk of vasospasm increases with each grade of the modified Fisher scale.
  grade 0: no visible SAH or intraventricular hemorrhage (IVH) grade 1: thin SAH, no IVH, grade 2: thin focal or diffuse SAH with IVH grade 3: thick focal or diffuse SAH without IVH grade 4: thick focal or diffuse SAH, IVH present
  units on a scale | 3.9 (.32) | 3.7 (.71) | 3.8 (.54)
Glasgow Coma Scale at Randomization [Mean (Standard Deviation); unit: units on a scale] — The Glasgow coma scale is used to assess responsiveness. The initial score correlates with the severity of brain injury and prognosis. The Glasgow Coma Scale provides a score in the range 3-15 and the sum of eye opening, motor and verbal responses. A higher score indicates less severe brain injury.
  units on a scale | 13.3 (2.7) | 10.7 (3.6) | 12.1 (3.3)
Location of Aneurysm [Count of Participants; unit: Participants]
  Anterior Cerebral Artery/Branches | 4 | 2 | 6
  Middle Cerebral/Internal Carotid Artery/Branches | 3 | 4 | 7
  Posterior Cerebral Artery/Branches | 1 | 0 | 1
  Vertebrobasilar System | 2 | 3 | 5
Treatment of Aneursym [Count of Participants; unit: Participants]
  Craniotomy | 4 | 2 | 6
  Endovascular | 6 | 6 | 12
  Unsecured | 0 | 1 | 1
Baseline Aspartate Aminotransferase [Mean (Standard Deviation); unit: units/liter] | 22.7 (5.7) | 25.5 (11.8) | 24.1 (9.0)
Baseline Aanine Transaminase [Mean (Standard Deviation); unit: units/liter] | 27.5 (13.4) | 24.4 (15.7) | 26.1 (14.2)
Baseline QTc Interval [Mean (Standard Deviation); unit: milliseconds] | 451.5 (24.3) | 456.4 (31.5) | 453.2 (27.0)
Admitted Intubated [Count of Participants; unit: Participants] | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events
Description: Summary tables and listings will be provided for all reported adverse events, defined as adverse events that start on or after the first administration of study drug. The reported adverse event term will be assigned a standardized preferred term.
  Adverse events will be summarized based on the number and percentage of patients experiencing the event. In the event a patient experiences repeat episodes of the same adverse event, then the event with the highest severity grade and strongest causal relationship to study treatment will be used for purposes of incidence tabulations.
  All deaths will be reported in a patient listing, which will include the primary cause of death and the number of days between the date of the last dose of study drug and death.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
Participants
  Venous Thromboembolism | 2 | 0
  Myocardial Infarction | 0 | 0
  Seizure | 1 | 1
  Any Documented Infection | 4 | 6
  Cerebral Salt Wasting | 3 | 2
  Leukopenia | 0 | 1
  Aneurysm Rebleed | 0 | 1
  Acute Respiratory Distress Syndrome | 0 | 1
  Death | 0 | 1

2. Secondary Outcome: Study Day 7 and Study Day 10 Serum and CSF EET/ Dihyroxyeicosatrienoic (DHET) Ratio, by Mass Spectroscopic Analysis (ng/mL)
Description: Day 7 and day 10 serum EET/DHET ratios will be measured by liquid chromatography and mass spectroscopy of collected blood samples.
  Day 7 and day 10 CSF EET/DHET ratios will be measured by liquid chromatography and mass spectroscopy of collected CSF samples.
Time Frame: 10 days
Population: Missing data occurred due to no sample collection from the CSF in patients who had external ventricular drains removed as part of their standard ICU care, prior to the study visit for sample collection. Missing serum samples are the result of one patient in the placebo group who died prior to sample collection visit, and multiple unsuccessful attempts at blood collection from another patient.
Measure: Mean (Standard Deviation); unit: ration
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
ration
  Study day 7 CSF 14,15-EET/DHET ratio: number analyzed (Participants) | 10 | 8
  Study day 7 CSF 14,15-EET/DHET ratio | .17 (.07) | .19 (.16)
  Study day 10 CSF 14,15-EET/DHET ratio: number analyzed (Participants) | 8 | 7
  Study day 10 CSF 14,15-EET/DHET ratio | .45 (.78) | .52 (1.04)
  Study day 7 serum 14,15-EET/DHET ratio | .30 (.11) | .12 (.03)
  Study day 10 serum 14,15-EET/DHET ratio: number analyzed (Participants) | 10 | 7
  Study day 10 serum 14,15-EET/DHET ratio | .27 (.07) | .12 (.02)

3. Secondary Outcome: Study Day 7 and Study Day 10 Serum Epoxyoctadecenoic Acid (EPOME) to Dihydroxyoctadec-12-enoic Acid (DPOME) Ratio, by Mass Spectroscopic Analysis (ng/mL)
Description: Study day 7 and study day 10 serum epoxyoctadecenoic acid (EPOME) to dihydroxyoctadec-12-enoic acid (DPOME) ratio, will be measure by mass spectroscopic analysis of collected blood samples.
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ration
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
ration
  Day 7 serum 12,13 EpOME/DiHOME ratio | 6.0 (4.3) | 1.8 (.92)
  Day 10 serum 12,13 EpOME/DiHOME ratio: number analyzed (Participants) | 10 | 7
  Day 10 serum 12,13 EpOME/DiHOME ratio | 8.7 (7.1) | 1.7 (.90)

4. Secondary Outcome: Serum Biomarkers of Endothelial Injury From Blood Samples Obtained on Study Day 7 and Study Day 10
Description: The following serum biomarkers will be obtained from collected blood samples by Luminex assay: e-selectin, p-selectin, Vascular cell adhesion marker (VCAM-1), Platelet endothelial cell adhesion marker (PECAM-1, CD31), intercellular adhesion molecule (ICAM-1).
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
ng/mL
  Serum Day 7 ICAM | 8.4 (7.5) | 8.3 (6.8)
  Serum Day 10 ICAM: number analyzed (Participants) | 10 | 7
  Serum Day 10 ICAM | 17.8 (27) | 6.7 (6.6)
  Serum Day 7 VCAM | 8.3 (3.0) | 7.9 (2.0)
  Serum Day 10 VCAM: number analyzed (Participants) | 10 | 7
  Serum Day 10 VCAM | 8.9 (2.9) | 7.9 (2.1)
  Serum Day 7 PECAM-1 | 1.4 (.56) | 1.7 (.90)
  Serum Day 10 PECAM-1: number analyzed (Participants) | 10 | 7
  Serum Day 10 PECAM-1 | 1.7 (.90) | 1.6 (.65)
  Serum Day 7 E-Selectin | 46.6 (25.3) | 48.0 (33.0)
  Serum Day 10 E-Selectin: number analyzed (Participants) | 10 | 7
  Serum Day 10 E-Selectin | 53.0 (23.8) | 44.7 (30.3)
  Serum Day 7 P-Selectin | 1.4 (.83) | 1.1 (.28)
  Serum Day 10 P-Selectin: number analyzed (Participants) | 10 | 7
  Serum Day 10 P-Selectin | 1.7 (.90) | 2.0 (2.2)

5. Secondary Outcome: CSF Biomarkers of Neuroinflammation, From Blood Samples Obtained on Study Day 7 and Study Day 10
Description: The following CSF biomarker will be obtained from collected CSF samples by Luminex assay: Tumor necrosis factor alpha (TNF-α) (pg/mL), Interleukin 1β (IL-1β) (pg/mL), Interferon gamma (IFN-γ) (pg/mL), Interleukin 6 (IL-6) (pg/mL), Interleukin 8 (IL-8) (pg/mL), Monocyte chemoattractant protein 1 (MCP-1) (pg/mL)
Time Frame: 10 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg / mL
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
pg / mL
  CSF Day 7 IFN-gamma: number analyzed (Participants) | 10 | 8
  CSF Day 7 IFN-gamma | 1.9 (1.0) | 4.6 (6.8)
  CSF Day 10 IFN-gamma: number analyzed (Participants) | 8 | 7
  CSF Day 10 IFN-gamma | 1.5 (.84) | 5.8 (12.9)
  CSF Day 7 IL-1b: number analyzed (Participants) | 10 | 8
  CSF Day 7 IL-1b | 1.6 (.82) | 5.0 (9.6)
  CSF Day 10 IL-1b: number analyzed (Participants) | 8 | 7
  CSF Day 10 IL-1b | 1.0 (.50) | 4.4 (9.2)
  CSF Day 7 IL-6: number analyzed (Participants) | 10 | 8
  CSF Day 7 IL-6 | 2991.2 (3420.0) | 3417.9 (4110.2)
  CSF Day 10 IL-6: number analyzed (Participants) | 8 | 7
  CSF Day 10 IL-6 | 2089.4 (3248.4) | 2051.6 (3570.7)
  CSF Day 7 IL-8: number analyzed (Participants) | 10 | 8
  CSF Day 7 IL-8 | 1652.4 (1374.4) | 3971.0 (3298.9)
  CSF Day 10 IL-8: number analyzed (Participants) | 8 | 7
  CSF Day 10 IL-8 | 1093.6 (775.3) | 1485.8 (1002.2)
  CSF Day 7 TNF-alpha: number analyzed (Participants) | 10 | 8
  CSF Day 7 TNF-alpha | 7.8 (2.6) | 13.1 (15.6)
  CSF Day 10 TNF-alpha: number analyzed (Participants) | 8 | 7
  CSF Day 10 TNF-alpha | 5.9 (2.8) | 8.1 (9.9)

6. Other Pre Specified Outcome: Hospital Length of Stay in Days
Description: The hospital length of stay will be recorded in days, at the time of hospital discharge.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
days | 16.9 (3.3) | 28.8 (19.8)

7. Other Pre Specified Outcome: Discharge Disposition
Description: The disposition from the hospital in one of the following categories: home, home with services, rehab, long term acute care facility, skilled nursing facility, hospice, death
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
Participants
  Discharged to home | 7 | 2
  Discharged to rehab, long term acute care facility, skilled nursing facility, hospice, death | 3 | 7

8. Other Pre Specified Outcome: Number of Participants With New Stroke on Hospital Discharge Imaging
Description: The last head CT or other brain imaging to detect the presence of a new area of cerebral infarction will be reviewed at the time of hospital discharge. A cerebral infarction will be defined as a one identified on hospital discharge that was not present on imaging between 24-48 hours after aneurysm occlusion, and not attributable to other causes such as surgical clipping or endovascular treatment. Hypodensities resulting from extraventricular drains or residual intraparencyhmal hematomas will not be considered new strokes.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
Participants | 1 | 1

9. Other Pre Specified Outcome: Modified Rankin Scale (mRS) at Hospital Discharge and 90 Day Follow up
Description: The mRS score will be determined by patient or surrogate interview, at both hospital discharge and 90 day follow up. Scores will be assigned based on the following: 0 - no symptoms, 1 - no significant disability, able to carry out all usual activities despite some symptoms, 2 - slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities, 3 - moderate disability, requires some help, but able to walk unassisted, 4 - moderately severe disability, unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5 - severe disability, requires constant nursing care and attention, bedridden, incontinent, 6 - deceased.
Time Frame: 90 days
Population: One subject in GSK2256294 group lost to followup
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale
  Hospital Discharge mRS | 3.4 (1.5) | 4.1 (1.4)
  90 day follow-up mRS: number analyzed (Participants) | 9 | 9
  90 day follow-up mRS | 2.2 (1.6) | 3.3 (1.7)

10. Other Pre Specified Outcome: Extended Glasgow Outcome Scale (GOSE) Score at 90 Day Follow up
Description: At 90 day follow up, the GOSE will be determined by patient or surrogate telephone interview, based on a structured interview of 19 questions. The GOSE is a scale of 1-8 where 1 - deceased, 2 - vegetative state, 3 - low severe disability, 4 - upper severe disability, 5 - low moderate disability, 6 -upper moderate disability, 7 - low good recovery, 8 - upper good recovery.
Time Frame: 90 days
Population: Missing data due to one subject in the GSK2256294 lost to followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GSK2256294 | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale | 5.4 (2.4) | 4.1 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 90 days after hospital discharge at the time of followup phone visit
Arm/Group | GSK2256294 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/9
Serious Adverse Events (participants affected / at risk) | 4/10 | 5/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2256294 (N=10) | Placebo (N=9)
Delayed Cerebral Ischemia (Nervous system disorders) | 2 (2) | 1 (1)
Rebleed of Unsecured Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Central Line Associated Bloodstream Infection (Infections and infestations) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pseudomonas Ventriculitis, Bacteremia, Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT03318783/Prot_SAP_000.pdf